CLINICAL TRIAL: NCT05503329
Title: Prognostic Value of Systemic Arterial Lactate Levels in Patients With ST-segment Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention
Brief Title: Prognostic Value of Lactate Levels in Patients With STEMI Undergoing Primary PCI
Status: Completed | Type: Observational
Sponsor: Ahmed Maher Teaching Hospital (Other Government)
Responsible Party: Principal Investigator, Ahmed Hamdy Abdelhasseeb, clinical doctor, Ahmed Maher Teaching Hospital
Other Study IDs: FWA000017585
Record Dates: First submitted 2022-08-14; First posted 2022-08-16 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: arterial lactate level — an arterial lactate level measured from arterial sample from STEMI patients

SUMMARY:
To assess the prognostic value of systemic arterial lactate levels in patients with ST segment elevation myocardial infarction undergoing primary PCI and correlate with the results of primary PCI and 30 days MACE follow up.

DETAILED DESCRIPTION:
* Study Population: STEMI patients treated with primary PCI.
* Study period: over 6 months.
* Sample Size: 300 patients.

All patients received the standard care for acute STEMI patients which is the primary percutaneous intervention in addition to medications.

Hyperlactemia is defined as elevated lactic acid level in the blood. The normal blood lactate level is (0.5-1 mmol/L).

All subjects were subjected to

1. Careful history taking
2. Full cardiac examination
3. Investigations include:

   1. 12 lead surface ECG.
   2. Lactate level and full labs
   3. Pre-discharge echocardiography
   4. Peri-procedural details of primary PCI

the investigators assessed the relation between hyperlactemia and coronary flow, peak cardiac enzymes, hemodynamic parameters and MACE in 30 days follow up

ELIGIBILITY:
Inclusion Criteria:

* Patient with ST-segment elevation myocardial infarction for the first time.
* Patients undergoing primary PCI.
* Adult patients ≥ 18 years old.

Exclusion criteria:

* Hemodynamically unstable patients.
* Patients with renal impairment (creatinine clearance < 30 ml/min).
* Patients who developed flow limiting coronary dissection or mechanical complication during the procedure.
* Patients presenting > 24 hours after symptoms onset.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: STEMI patients treated with primary PCI
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Major adverse caediac events | 30 days
  we follow up occurrence of death, reinfarction, repeated hospitalization and new onset heart failure

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Maher teaching hospiral, Cairo, Elsayda Zainab Square, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdel-Salam A, El-Sayed A, Abdel-Haseeb A, Ibrahim M. Prognostic value of arterial lactate index in ST-elevation myocardial infarction treated with primary percutaneous coronary intervention: a prospective cohort study. Future Cardiol. 2023 Dec;19(16):767-777. doi: 10.2217/fca-2023-0065. Epub 2023 Dec 21. PMID 38127545